CLINICAL TRIAL: NCT05555823
Title: A Phase I Dose Escalation Study of Ascending Single and Multiple Doses of the MEK Inhibitor Zapnometinib in Healthy Subjects to Evaluate the Safety & Tolerability Compared to Placebo, Additionally Evaluating Pharmacokinetics and Pharmacodynamics of Target Engagement, as Well as Investigating Possible FDI and DDI
Brief Title: Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, Food Effect and DDI of Ascending Doses of the MEK Inhibitor Zapnometinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atriva Therapeutics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ATR-002-102
Record Dates: First submitted 2022-09-13; First posted 2022-09-27 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Healthy
MeSH Terms: interventions — 2-(2-chloro-4-iodophenylamino)-N-3,4-difluorobenzoic acid; repaglinide; Celecoxib

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, mono-centre; SAD, MAD, FDI, DDI part
Who Masked: Participant, Investigator
Masking Description: matching placebo tablets
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: ATR-002 (Experimental): In the SAD part, study participants will receive IMP orally once (except for the first cohort), or twice (two single doses separated by an adequate washout period of at least 10 days for the FDI cohort, which will be conducted according to a two-period fixed-sequence design with all subjects receiving the treatment sequence 'fasted-fed'). In each of the periods of the MAD Part, study participants will receive the IMP for seven consecutive days. Dosing will start at 600 mg (SAD part) and 900 mg (MAD part) in the first cohort and follow the dose escalation schedule that is given in the study protocol.
  Interventions: Drug: ATR-002
- Placebo Comparator: Placebo (Placebo Comparator): In the SAD part, study participants will receive IMP orally once (except for the first cohort), or twice (two single doses separated by an adequate washout period of at least 10 days for the FDI cohort, which will be conducted according to a two-period fixed-sequence design with all subjects receiving the treatment sequence 'fasted-fed'). In each of the periods of the MAD Part, study participants will receive the IMP for seven consecutive days.
  In the DDI period with repaglinide two doses of ATR-002 will be given, and in the DDI period with celecoxib, four doses of ATR-002 will be given.
  Interventions: Drug: Placebo; Drug: Repaglinide; Drug: Celecoxib

INTERVENTIONS:
Drug: ATR-002 — 300 mg tablets for oral intake
  Other Names: Zapnometinib
  Arms: Experimental: ATR-002
Drug: Placebo — matching tablets for oral intake
  Arms: Placebo Comparator: Placebo
Drug: Repaglinide — 0,5 mg tablets for oral intake
  Other Names: Repaglinide-ratiopharm
  Arms: Placebo Comparator: Placebo
Drug: Celecoxib — 100 mg capsules for oral intake
  Other Names: CELEBREX
  Arms: Placebo Comparator: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of ascending doses of the MEK-inhibitor zapnometinib (ATR-002) given as single doses (SAD Part) and as multiple doses for 7 days (MAD Part) in healthy subjects.

DETAILED DESCRIPTION:
This is a Phase 1, single-center, randomized, double-blind, controlled clinical trial (zapnometinib vs. placebo in the SAD/MAD Parts; 'fed' vs. 'fasted' in the FDI Part, 'probe substance' (repaglinide or celecoxib) in combination with zapnometinib vs. probe substance alone in the DDI part). The study will assess the safety, tolerability, PK (applicable to SAD/MAD Part) and PD (applicable to SAD Part only) effects of zapnometinib versus a matching placebo (applicable to SAD/MAD Part) in healthy subjects. The FDI cohorts will investigate the possible impact of a standard breakfast high in fat content in comparison to administration in fasted state. The DDI cohorts with celecoxib and repaglinide will investigate a possible drug-drug interaction.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent as described in Section 10.1.3, which includes compliance with the requirements, prohibitions and restrictions listed in the informed consent form (ICF) and in this protocol.
2. Subject has been informed both verbally and in writing about the objectives of the clinical trial, the methods, the anticipated benefits and potential risks and the discomfort to which he/she may be exposed, and has given written consent to participation in the trial prior to trial start and any trial-related procedure.
3. Study participant must be at least 18 years of age and not older than 55 years of age at the time of signing the ICF.
4. Non-smokers or ex-smokers who had stopped smoking for at least 5 years prior to start of the clinical study.
5. In good physical and mental health as determined on the basis of medical history and general physical examination performed at screening.
6. Hematology and chemistry parameters, pulse rate and/or blood pressure, and ECG within the reference range for the population studies, or showing no clinically relevant deviations, as judged by the Investigator (Note that some defined clinical laboratory parameters must not exceed the upper limit of reference range - see Exclusion Criterion #3).
7. Negative urine test for selected drugs of abuse at screening and upon check-in at the clinical site. Note: Subjects should not consume poppy-seeds within 72 h before screening and before each urine drug screening because this can falsify the results of the opiate urine drug test.
8. Negative alcohol breath test at screening and upon check-in at the clinical site.
9. Negative hepatitis panel (including hepatitis B surface antigen [HBsAg] and anti-hepatitis C virus [HCV] antibodies) and negative human immunodeficiency virus (HIV) antibody screens and negative SARS-CoV-2 PCR test.
10. Body weight at least 70 kg for males and 60 kg for females and have a body mass index (BMI) ≥ 18.0 kg/m2 and < 29.9 kg/m2.
11. Male or female. Pregnancy and Contraception
12. Female subjects must be of non-childbearing potential, as follows.

A female study participant is eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies:

1. At least 1 year post-menopausal (amenorrhea >12 months in the absence of an alternative medical cause and follicle-stimulating hormone >30 mIU/mL in women not using hormonal contraception or hormonal replacement therapy) prior to screening;
2. Surgically sterile (bilateral oophorectomy, hysterectomy, bilateral salpingectomy, or bilateral tubal ligation).

To protect partners from possible exposure to study medication in semen, male subjects must use a condom during the study, even if they have had a vasectomy or their partner is not of childbearing potential, and they must not plan to father a child, or donate sperm, during the study, and for 4 months after their final dose of study medication. Note: medically acceptable methods of contraception that may be used by the partner include combined oral contraceptive, contraceptive vaginal ring, contraceptive injection, intrauterine device, and etonogestrel implant.

Exclusion Criteria:

1. Clinically relevant abnormal history, physical findings, ECG, or laboratory values at the pre-study screening assessment that could interfere with the objectives of the study or the safety of the subject. Note: Blood pressure and heart rate at the screening examination outside the ranges 90- 139 mmHg systolic, 50-89 mmHg diastolic; heart rate 50-90 bpm are considered as exclusion criteria.
2. QTc interval of ECG above the upper limit of reference range at screening. The following commonly accepted reference range will be taken as a basis: Men: QTc ≤ 440 ms; Women: QTc ≤ 460 ms.
3. Aspartate aminotransferase [AST], alanine aminotransferase [ALT], alkaline phosphatase [AP], glutamate dehydrogenase [GLDH], gamma glutamyl transpeptidase [γ-GT]) above the upper limit of the reference range.
4. Presence of acute or chronic illness or history of chronic illness sufficient to invalidate the subject's participation in the study or make it unnecessarily hazardous.
5. A condition that, in the opinion of the Investigator, could compromise the well-being of the subject or course of the study, or prevent the subject from meeting or performing any study requirements.
6. Impaired endocrine, thyroid, hepatic, respiratory or renal function, diabetes mellitus, coronary heart disease, cancer, or history of any psychotic mental illness.
7. Respiratory tract infection within 4 weeks before the screening visit.
8. History of surgery or medical intervention, or planned surgery or medical intervention, that could interfere with the objectives of the study or the safety of the subject.
9. Presence or history of severe adverse reaction to any drug, or sensitivity to components of the study medication.
10. Loss of more than 400 mL blood, e.g., as a blood donor, or donation of blood products, during the 3 months before the study.
11. Positive fecal blood test at screening.
12. Active or latent parasitic infection, visit to a country with a high prevalence of parasitic infections within 3 months before receiving study medication.
13. Use of any prescription or over-the-counter medicine, with the exception of acetaminophen (paracetamol), within 14 days (or 5 half-lives, whichever is longer) before the first dose of study medication as defined in Section 10.5.
14. Treatment with any known enzyme inducing or inhibiting agents (e.g., St. John's Wort (Johanniskraut), barbiturates, phenothiazines, cimetidine, ketoconazole etc.) within 30 days before first administration of IMP or during the trial.
15. Presence or history of drug or alcohol abuse, or intake of more than 21 units (14 units for women) of alcohol weekly.
16. Receipt of a living vaccine within the 3 months, or mRNA or vector vaccine against COVID-19 within 4 weeks before dosing, or planned vaccination during the study.
17. Currently participating in other clinical trials or previous treatment with an investigational medicinal product within 5 half-lives or 30 days (whichever is longer) prior to randomization.
18. Known allergy or hypersensitivity to the IMP (including excipients) or history of severe adverse reaction to any drug, or sensitivity to components of the study medication.
19. Study participant is pregnant or breastfeeding.
20. Subject has been committed to an institution by virtue of an order issued either by the judicial or the administrative authorities.
21. Subject is an employee of the sponsor, or an employee of any third-party organization involved into the clinical trial, or an employee of the clinical trial site, or is dependent on the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with TEAEs and SAEs, with abnormal ECG readings, abnormal vital signs, and abnormal laboratory parameters | From 1st administration of study drug (SAD/MAD Day 1; DDI Day -1) up to 21 days after last dosing

SECONDARY OUTCOMES:
SAD part: Cmax | Day 1 to Day 7
SAD part: tmax | Day 1 to Day 7
SAD part: t1/2 | Day 1 to Day 7
SAD part: AUC0-t | Day 1 to Day 7
SAD part: AUC0-∞ | Day 1 to Day 7
MAD part: Cmax | postdose on Day 1
MAD part: tmax | postdose on Day 1
MAD part: Ctrough | Day 2 to Day 7
MAD part: Cmax | postdose on Day 7
MAD part: tmax | postdose on Day 7
MAD part: t1/2 | postdose on Day 7
MAD part: AUC0-t | postdose on Day 7
SAD part: percent MEK inhibition by measuring the reduction of ERK phosphorylation after study drug administration as compared to baseline in stimulated PBMCs isolated from blood samples from study participants | up to day 5
FDI cohort (two-period fixed-sequence design 'fasted' vs. 'fed'): Cmax | Day 1 to Day 7
FDI cohort (two-period fixed-sequence design 'fasted' vs. 'fed'): tmax | Day 1 to Day 7
FDI cohort (two-period fixed-sequence design 'fasted' vs. 'fed'): t1/2 | Day 1 to Day 7
FDI cohort (two-period fixed-sequence design 'fasted' vs. 'fed'): AUC0-t | Day 1 to Day 7
FDI cohort (two-period fixed-sequence design 'fasted' vs. 'fed'): AUC0-∞ | Day 1 to Day 7
DDI part: Cmax | Day -1 and Day 1
DDI part: tmax | Day -1 and Day 1
DDI part: t1/2 | Day -1 and Day 1
DDI part: AUC0-t | Day -1 and Day 1
DDI part: AUC0-∞ | Day -1 and Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Atriva study site, Neu-Ulm, Germany